# IMPACT OF A PHARMACEUTICAL INTERVENTION TO IMPROVE ADHERENCE OF INHALED MEDICATION IN ASTHMA AND COPD PATIENTS: STUDY PROTOCOL FOR A RANDOMIZED CONTROLLED TRIAL

Claudia Gregoriano<sup>1,2</sup>, Thomas Dieterle<sup>1,3</sup>, Selina Dürr<sup>1</sup>, Isabelle Arnet<sup>2</sup>, Kurt E. Hersberger<sup>2</sup>, Jörg D. Leuppi<sup>1,3</sup>

<sup>1</sup> University Clinic of Medicine, Cantonal Hospital Baselland, Liestal, Switzerland.

<sup>2</sup> Department of Pharmaceutical Sciences, University of Basel, Switzerland

<sup>3</sup> Faculty of Medicine, University of Basel, Basel, Switzerland

#### Corresponding author:

Claudia Gregoriano

University Clinic of Medicine, Cantonal Hospital Baselland

Rheinstrasse 26, Liestal CH - 4410, Switzerland

Phone: +4161 925'37'65

Fax: +4161 925'28'83

Email: claudia.gregoriano@ksbl.ch

Document Date: 04. February 2017

Word count (excluding title page, abstract, references, figures and tables): 3'979 words

# **ABSTRACT**

**Introduction**: Despite progress in pharmacological and non-pharmacological treatment in recent years, the burden of disease among asthma and COPD patients is high and patients may be frequently hospitalized due to exacerbations. Reasons for uncontrolled disease are manifold, but are frequently associated with poor inhalation technique and non-adherence to the prescribed treatment plan which may cause substantial mortality, morbidity, and cost to the healthcare system. In this respect, the study of causes for non-adherence and the development of measures to increase respectively maintain treatment adherence, particularly in chronic diseases, is of major clinical importance.

Therefore, the primary aim of this study is to measure medication adherence in patients with chronic obstructive lung diseases such as asthma and COPD, and to investigate the impact of a reminder on disease outcomes and quality of life.

Methods and analysis: In this ongoing prospective single-blind randomized controlled study, the adherence to inhaled medication is analyzed over a six-months period in in- and outpatients with asthma or COPD, who have experienced at least one exacerbation during the last year. Adherence is measured using electronic data capture devices which save date and time of each inhalative device actuation and transfer these data daily via wireless-connection to a web-based database. Patients are randomly assigned to an intervention, respectively control group. Patients assigned to the intervention group will receive audio reminder and support calls in case medication is not been taken as prescribed or if rescue medication is used more frequently than prespecified in the study protocol. During the study, participants are assessed every two months.

**Ethics and dissemination:** The study has been approved by the Ethics Committee of Nordwest- and Zentralschweiz (registry number: EK- 269/13). The results of this study will be disseminated via scientific seminar and conference presentations and in academic peer-reviewed journals.

**Trial registration:** ClinicalTrials.gov: NCT02386722.

## STRENGTHS AND LIMITATIONS OF THIS STUDY

- Adherence estimation using state of the art method
- The primary outcome is of clinical relevance
- Primarily real-life study setting
- A limitation of this study is that we have a potential selection bias
- Single-centre and not multi-centre study

# Introduction

Asthma and chronic obstructive pulmonary disease (COPD) are both prevalent lung diseases that require daily and often lifelong-use of inhaled medication[1]. According to the World Health Organisation (WHO) COPD currently represents the fourth leading cause of death worldwide and is predicted to become the third leading cause of death by 2030[2]. The prevalence of COPD is increasing due to continuing exposure to COPD risk factors (i.e. tobacco smoke or air pollution) and the continuously aging world's population[3]. The prevalence of asthma is increasing as well[4]. In Swiss adults, prevalence of asthma and COPD was found to be around 7% and 7-9%, respectively[5, 6].

### TREATMENT AND DISEASES CONTROL

Despite progress in pharmacological and non-pharmacological treatment in recent years, the burden of disease among asthma and COPD patients is high and patients may be frequently hospitalised due to exacerbation. Based on data from the Swiss COPD cohort, the exacerbation rate is 23% per year[7]. Acute exacerbations are a risk factor for disease progression, and are associated with higher mortality[8]. A survey published by Leuppi et al. showed that the level of asthma control in Switzerland is very low with 15% of all the investigated patients[9]. This has also been confirmed by a cross-sectional survey of Miedinger et al. that found controlled asthma in 27% of all patients according to the international GINA guidelines[10]. A good adherence to therapy can increase the likelihood of achieving better asthma control[11].

Reasons for lack of diseases control in asthma and COPD are manifold, but are frequently associated with poor inhalation technique and non-adherence to prescribed treatment plan, which may influence diseases' mortality and morbidity as well as the costs to the health care system[12].

#### MEDICATION ADHERENCE

According to WHO, adherence is defined as "the extent to which a person's behaviour (including medication-taking) corresponds with agreed recommendations from a health care provider"[13]. Adherence represents the basic condition for the effectiveness of drug therapy and for complete disease control. Non-adherence not only leads to suboptimal treatment of individual patients. It also causes disease prolongation and increases hospital readmissions what in turn leads to an increase of the health care system costs[14].

Based on a systematic review of medication adherence literature, Vrijens et al. proposed a new taxonomy for describing and defining adherence to medication[15]. The Ascertaining Barriers to Compliance (ABC) taxonomy considers a sequence of events that have to occur for a patient to achieve an optimal benefit from his or her prescribed treatment regimen and to minimize the risk of harm. This process is divided into 3 essential components, which are

initiation, implementation and persistence. The process starts with the initiation, characterised by the intake of the first dose of a prescribed medication by the patients. It continues with the implementation of the dosing regimen, which is defined as the extent to which a patient's actual dosing corresponds to the prescribed medication, from initiation until the last dose is taken. This represents a longitudinal description of patient behaviour over time. The last step of the process is the persistence, which is the time duration from initiation, until eventual treatment discontinuation. After discontinuation, a period of nonpersistence may follow until the end of the prescribed period.

According to the above defined processes, non-adherence to medications can occur in the following situations: late or non-initiation of the prescribed treatment, suboptimal implementation of the dosing regimen or early discontinuation of the treatment. The subdivision into individual processes helps to focus research questions and to find measures and corresponding data to answer them.

On average, adherence to long-term therapy is estimated to be around 50% as shown in a systematic review summarising the results of randomised controlled trials (RCTs) of interventions to help patients follow prescriptions for medications for medical problems[16]. In general, adherence to medication can be measured using direct or indirect methods. Direct methods include direct observation of drug intake or measurement of drug concentration respectively biologic markers in blood, urine, or other body fluids. Indirect methods include assessment of a patient's clinical response, pills count, rates of refilling prescriptions, patient's self-report, and as most recommended method the electronic monitoring[17, 18]. Currently, no method is considered to represent the gold standard for measuring adherence to medications[19, 20]. Nevertheless, the method of choice that has emerged recently is the use of electronic monitoring[21].

A review by Makela et al.[22] analysed studies about asthma and COPD adherence between 2000 and 2012. The three leading methods were self-reported measures (37.8%), prescription refill adherence (32.8%) and electronic monitoring (19.1%)[22].

Self-reporting by patients was shown to be the most cost-effective in clinical and research settings[22]. However-being a subjective method-it also bears the highest risk of overestimating adherence compared to electronic measurements[23].

Observational retrospective studies based on dispensing data from pharmacy record database analyzed the refill adherence for different inhaled medication in asthma and COPD patients[24-26]. The importance of refill adherence is limited, since this measurement cannot assess the timing of the ingested or inhaled doses, which depends on the duration of drug action, and this has an important impact on the efficacy of treatment[27].

To investigate the variability in timing and taking adherence, measurements of dose and timing are necessary, which can be done with electronic medication monitors. Electronic monitoring provides precise data on the timing and pattern of inhaler actuation as well as detect multiple successive actuations (dumping)[28]. Electronic monitoring methods are non-invasive and represent one of the best ways to detect adherence patterns when using additional tools attached on the inhaler devices[29]. One of the electronic monitoring systems on the market are SmartInhaler<sup>TM</sup> devices (Adherium Ltd., Auckland, New Zealand), which have been validated for the assessment of adherence to inhaled medication on a daily basis[30]. The SmartInhaler<sup>TM</sup> devices are able to track time and date of each actuation of the inhaler device (incorporated switch activates by depression or rotation of the device) and

transmit the data via a wireless connection to a secure web database[30]. This method of electronic monitoring has been used in several studies measuring adherence to inhaled medication[31, 32]. One study conducted with asthma patients using inhalative corticosteroids showed that the integrated audio-visual reminder function of these devices significantly improved adherence to inhaled medication[33]. For orally administered drugs or inhaled medications available as powder capsules, a new technology is used, which is called Polymedication Electronic Monitoring System (POEMS). This technology is composed of printed electronics, self-adhesive polymer film carrying loops of conductive wires that can be affixed to multidose punch card (Pharmis GmbH, Beinwil am See, Switzerland) with 28 cavities. Every time a powder capsule is taken out of the blister, a loop is broken leading to changes in electrical resistance that can be measured and recorded with date and time[34]. The reports generated by Smartinhalers and POEMS allow to detect whether the patients have taken the medication at the right time and dose.

#### INTERVENTIONS TO IMPROVE MEDICATION ADHERENCE

Maintenance of a sufficient adherence to the prescribed medication is of major importance for achieving a therapeutic success, particularly in chronic diseases. Haynes et al.[35] have reviewed randomized controlled intervention trials to improve the adherence to pharmacological regimens in patients with chronic diseases, including asthmatic patients. Both, adherence and clinical outcomes were measured in these studies. The authors found that less than 50% of the interventions achieved a significant improvement of adherence while only 30% demonstrated an improvement in clinical outcome. The best success was attained with interventions combining several intervention strategies (information, reminders, self-monitoring, reinforcement, counselling, telephone follow-up, supportive care, etc.). Interventions to improve medication adherence have had mixed results and successful interventions had been shown as usually complex[35].

#### STUDY OBJECTIVE

The objective of this study is to investigate the adherence to inhaled medication in asthma and COPD patients with an innovative methodology using specific electronic devices, which are able to provide data about the timing of inhaler action. Moreover, we want to assess the effect of an acoustic reminder and a close supervision by a pharmacist on the adherence, course of diseases and quality of life.

# METHODS AND ANALYSIS

#### PARTICIPANTS AND RECRUITMENT

In- and outpatients with a diagnosis of asthma bronchiale or COPD from several hospitals in the Basel region illustrated on table 1 and patients treated by pulmonologists in private practice are screened for eligibility. In addition, advertisement is made using posters, flyers, as well as on ad-screens (Cantonal Hospital Baselland Liestal and Bruderholz) including the most important information about the study. Advertisement is also placed in local newspapers.

Table 1 Recruitment locations and related recruitment types

| _Hospital | Location | Type of recruitment |
|---|---|---|
| Cantonal Hospital Baselland | Liestal,<br>Switzerland | - Screening of hospitalized |

| | | patients - Screening of emergency department - Screening of DRG-lists |
|---|---|---|
| Cantonal Hospital Baselland | Bruderholz,<br>Switzerland | <ul><li>Screening of DRG-lists</li><li>Collaboration with pulmonology department</li></ul> |
| Claraspital | Basel,<br>Switzerland | <ul> <li>Collaboration with pulmonology<br/>department</li> </ul> |
| Clinic Barmelweid | Barmelweid,<br>Switzerland | <ul> <li>Collaboration with pulmonology<br/>department</li> </ul> |
| Gesundheitszentrum Fricktal AG | Rheinfelden,<br>Switzerland | <ul> <li>Collaboration with pulmonology<br/>department</li> </ul> |

DRG, Diagnosis Related Groups.

In- and exclusion criteria initially are checked via telephone or during hospitalizations or practice visits. Eligible patients are invited for an initial training course. Before the study start, the investigator provides written and verbal information on content and duration of the study. In case of willingness to participate, patients have to sign an informed consent.

#### PATIENT INCLUSION CRITERIA

- males and females aged ≥18 years with
- asthma- and/or COPD diagnoses and
- prescribed daily inhaled medication with
- at least one exacerbation in the previous twelve months

#### PATIENT EXCLUSION CRITERIA

- patients with malignancies and/or other severe diseases or
- insufficient German language
- pregnant or lactating women

Enrolment started on January 2014 and will end as soon as at least 154 individuals are included in the study.

# STUDY DESIGN AND PROCEDURES

In this prospective single-blinded randomized controlled trial (RCT) (see figure 1 for study flow chart) 169 participants are followed up for six months. Prior to study start, patients have to be in a stable phase of their obstructive lung disease, which is defined as an exacerbation-free period of at least one month prior to commencement of the study and no current hospitalization for any other medical condition. Study participants will continue to be cared by their usual treating physician(s). They decide on all prescriptions and treatments.

All participants take part in a training course before the baseline visit. The goal of the training course is to provide refresher training on inhalation techniques in order to ensure that all participants are at the same level of disease knowledge and use their medication correctly. The training begins with a brief introduction about asthma and COPD. Then, the most frequently used devices are presented and briefly demonstrated. Correct technique depends on inhaler type, and it is important that patients use their own inhaler correctly. In addition, common mistakes and problems associated with the use of the devices are explained. The

correct use of the individual devices is demonstrated by a short film (produces by the "Deutsche Atemwegsliga" Bad Lippspringe, Germany)[36] which presents the most important steps to follow in order to achieve an effective inhalation. Notably, it has been shown that the manufacturer's instruction sheet is not effective enough to achieve correct techniques[37-39]. In contrast verbal and visual instructions seem to have a higher success rate in improving the application of inhalation devices[40]. At the end of the training, participants are given the opportunity to ask questions concerning the devices.

Visits take place at baseline (T0), after two (T1), four (T2) and six months (T3). Each visit includes a spirometry (EasyOne Pro, ndd Medizintechnik AG, Zurich, Switzerland), measurement of diffusion capacity (EasyOne Pro, ndd Medizintechnik AG, Zurich, Switzerland), exhaled nitric oxide (NIOX MINO®, Aerocrine AB, Sweden) and carbon monoxide (piCO+ Smokerlyzer, Bedfont Scientific Ltd., Kent, UK) measurements. To detect false device applications, each patient is asked to demonstrate the inhalation technique with all prescribed devices to the investigator using a placebo device (to avoid overdosing). Moreover, participants have to fill out the COPD Assessment Test (CAT)[41], the Asthma Control Test (ACT)[42], the St. George's Respiratory Questionnaire (SGRQ) and the Short Form (SF)-36[43, 44] to assess quality of life at baseline, after two, four and six months. To assess patients' beliefs about the necessity of the prescribed medication and their concern about the potential adverse consequences of taking it, the Beliefs about medicines Questionnaire (BMQ) is used at baseline[45, 46]. During these visits we also obtain information about exacerbation since the previous visit.

#### RANDOMIZATION

After having given written informed consent eligible subjects are randomly assigned either to the intervention or to the control group. The intervention group is provided with an acoustic reminder for inhalation and receives support calls when the medication is not taken as prescribed while the control group receive no further support regarding the adherence. A randomization list with study group allocation is generated using R (RStudio®, Boston, USA). Randomization procedure is provided in block size of two. Therefore, examinations between study groups are sequent. This reduces the risk of a season effect between study groups. The patients are not aware of which group they have been randomized to (single-blinded).

#### **CLINICAL INTERVENTIONS**

Patients assigned to the intervention group receive an audio-reminder, generated by a smartphone. For patients with Smartinhaler, the inhalation times are entered on the Smartinhalerlive.com website by the investigator. These are generated by an app on the smartphone. For patients with POEMS, the inhalation times are entered also by the investigator directly as an alarm clock on the smartphone. Patients were allowed to choose the inhalation times themselves, depending on their personal habits and daily routine, and it was possible to define a time for the working days and a time for the weekend. In both cases, the generated reminders have to be stopped by the patient and will have no link to the inhalation actuation. Moreover, these patients receive support calls when the use of rescue medication doubles or if the inhaled medication is not inhaled as prescribed for more than two consecutive days. They also receive a feedback on their adherence at each visit, especially for the results of the POEMS.

Patients assigned to the control group have no reminder and will receive no further support regarding the adherence of their inhaled medication.

#### CALCULATION OF SAMPLE SIZE

"Time to next exacerbation" is subject to the power calculation. A previous study has shown that 30% of COPD patients are readmitted again within six months because of an exacerbation[47]. We expect that 12% of the patients in the intervention group will have an exacerbation. This corresponds to a hazard ratio (intervention/control) of 0.36. Assuming a sample size of 70 subjects for each study group, there is a power of 80% to detect a HR of 0.36 based on a one-tailed test. The calculation is based on the assumptions mentioned above and on a one-tailed significance level of 5%. Additional 14 subjects (7 for each study group) have been added to account for dropouts. Therefore, 154 subjects will be investigated in this study.

#### MEASUREMENT OF OBJECTIVE ADHERENCE

Adherence is measured in both groups using Smartinhalers and POEMS as outlined above. Daily measurements are started after the baseline visit (T0) and are continued until the end of the study (visit T3).

Recorded data are uploaded daily at 00:00 to a web-based database via a wireless connection. Participants are asked to take their medication at the first visit in order to ensure the correct handling and usage of the Smartinhaler. Once the devices are installed on the inhalers, patients can use their medication as usual.

Currently, no monitoring devices exist that were specifically developed for monitoring the adherence of the newly introduced inhalation-device Ellipta<sup>®</sup>. To assess adherence in patients undergoing treatment with Ellipta<sup>®</sup> a Smartinhaler with a placebo-device is handed out and patients are instructed to trigger a puff of the placebo every time when they inhale their active treatment. This procedure allows an indirect recording of date and time actuation of the Ellipta<sup>®</sup> inhaler.

For inhalation with powder capsules (Breezhaler and HandiHaler), POEMS are used. The capsules are pre-filled for the following 2 weeks with a patient's individualized prescription plan (mostly one time daily inhalation of capsule contents). The multidose punch cards are filled manually by a pharmacist. The participants with Breezhaler and HandiHaler will receive one multidose punch card for every 2 weeks. Every time the patients break a loop for taking the capsules, date and time are recorded on a microchip, which can be read when the patients bring back the empty punch card.

#### DATA COLLECTION AND OUTCOME MEASURES

The primary outcome of this study is "time to next asthma or COPD exacerbation", defined as acute-onset worsening of the patient's condition beyond day-to-day variations requiring interaction with a health care provider[48], which may occur during the index exacerbation or follow-up. Data collections about this outcome are assessed after two, four and six months (number of exacerbations since last visit with exact period of exacerbation and number of exacerbation with hospitalization). If patients are not able to give information about the time of exacerbation, treating physician is contacted.

Sociodemographic variables such as gender, civil status, age, education level and employment status are obtained by a generic questionnaire at the baseline visit. Furthermore, body mass index (BMI), smoking status, as well as pack years (py) are assessed during this visit. In addition, disease-related questions such as allergies,

comorbidities, current medication and number of exacerbations in the previous twelve months are recorded including hospitalizations and emergency department attendance.

This project focuses on the implementation of a prescribed dosing regimen. Objective adherence will be analyzed according to the following widely used definitions[49]:

- Taking adherence: (Number of puffs inhaled during 24h/number of puffs prescribed during 24h) x 100.
- Timing adherence: (Number of correct dosing intervals during 24 hours/number of dosing intervals during 24 hours) x100; correct dosing intervals are prescribed intervals ±25%:
  - o For once daily dosing: 24h±25%=18-30h
  - o For twice daily dosing: 12h±25%= 9-15h
  - o For three daily dosing: 8h±25%= 6-10h
- Gaps: (Number of days without inhalation during the whole study period/number of days in same time period) x 100.
- Maximal gap length: Number of consecutive days of the longest period of time without inhalation.

Different lung function tests are performed at baseline, after two, four and six months to assess changes in lung function (FEV<sub>1</sub>, FVC, FEV<sub>1</sub>/FVC), diffusion capacity, NO-measurements and CO-measurements.

To evaluate the inhalation technique, participants demonstrate at baseline and at every follow up visit how they actually use their device at home. For this purpose, placebo devices are used to prevent overdosing. Correctness of inhaler use is assessed using pre-defined checklists for each inhaler type based on user guidelines and instruction package inserts from the manufacturers[50-55]. Correct inhaler usage is defined as correct performance of every step on the checklist. Incorrect inhaler usage is defined as one or more steps done incorrectly. A total score is calculated (incorrect application =0, correct application =1) and applied to every step. Possible errors are corrected by verbal instruction and visual demonstration. For ethical reasons the correction was performed in both groups. Patients demonstrate their inhalation technique until it is performed correctly.

To assess patients' beliefs about the need of the prescribed medication and their concerns about the potential adverse consequences of taking it, the BMQ is used at baseline.

Changes in quality of life are assessed at baseline, after two, four, six months using different disease-specific questionnaires: SGRQ, CAT and ACT. To assess general quality of life, SF-36-questionnaire is used.

## STATISTICAL ANALYSIS

Statistical analyses, including descriptive statistic and survival analyses, are done using the software R (RStudio®, Boston, USA) and SPSS (IBM Corporation, Armonk, USA). Statistical significance is set at the 5% level. Time to next exacerbation is compared using the Kaplan-Meier method and Cox proportional hazard model. Results will be reported as HR (hazard ratio) with corresponding 95% confidence interval (CI) and p-value. A hazard ratio smaller than one is expected. This means that the intervention group will have a smaller risk for exacerbations. Associations between time to between exacerbation and independent predictors will be analyzed (taking adherence, timing adherence and gaps without

inhalation). Comparisons of secondary parameters are done using t-tests or chi-square-tests (or their nonparametric equivalents if continuous data are not normally distributed).

#### HANDLING OF MISSING DATA AND DROP OUTS

Patients will be rated as drop out when they will be excluded from the study at their request or if they will be no longer able to participate in the study until the final visit at six months. Patients, who will not be able to undergo all clinical examination during the follow-up visits, will remain in the study. Multiple imputation methods will be used to impute missing data with less than 25% missing values, which is typically more efficient than complete cases analysis when covariates have missing values[56].

#### **ETHICS AND DISSEMINATION**

This study is conducted according to the Helsinki Declaration and according to the good clinical practice guidelines. The study participation of the patients is voluntary and can be revoked at any time without specification of reasons and will have no disadvantages for their future medical care. The study was approved by the Ethics Committee of Nordwest- and Zentralschweiz (registry number: EK- 269/13) and was registered in the https://clincialtrials.gov/trials database (NCT02386722).The results of this study will be disseminated via seminar and conference presentations and in academic peer reviewed journals.

# DATA SECURITY/DISCLOSURE OF ORIGINAL DOCUMENTS

All patients' data are collected and stored under confidentiality rules. All study related data and documents are stored on a protected server of the Cantonal Hospital Baselland. Data access is limited to members of the Medical research group at the Cantonal Hospital Liestal. After the end of the study, all documents and informed consent are retained in the archive of the University Department of Internal Medicine at the Cantonal Hospital Liestal for 10 years according to the applicable Swiss regulatory requirements.

# EXPECTED RESULTS AND SIGNIFICANCE OF THE RESEARCH PROJECT

To date, only few studies have investigated medication adherence in patients with chronic obstructive lung diseases. These studies were retrospectively analysed and limited to refill adherence, comprising several important limitations, such as not assessing the relationship between the duration of drug action and the timing of the ingested doses, which has an important impact on the efficacy of treatment[57]. Other disadvantages of this measurement are missing data, if refill medication is obtained outside of the investigated system and incomplete records if the medication plan is verbally modified by the prescriber without informing the dispensing pharmacy. Moreover, assumptions have to be made on medication-taking behaviour corresponding to prescription refilling and the medications that are taken according to prescription[58].

We expect that a regular adherence reminder and a close supervision by a health care professional will have a beneficial effect on the adherence to inhaled medication in patients with asthma or COPD, resulting in an increased time to next exacerbation. Moreover, we expect that an improved adherence will increase the quality of life in these patients.

With the prospective study design and the use of state-of-the-art devices for measuring adherence, we expect scientifically relevant and clinically meaningful results that will have a

substantial and positive impact on the provision of health care in chronically ill patients with asthma or COPD.

# **CONTRIBUTORS**

CG TD and JDL are chief investigators of the project. CG, TD, SD, IA, KH and JDL made contributions to the protocol in their specific areas of expertise. CG prepared the first draft of this manuscript and all authors revised the paper critically for important intellectual content and gave approval for the final version.

# **FUNDING**

This project is financially supported by grants from the Gottfried und Julia Bangerter-Rhyner Foundation, Bern, Switzerland, and the Swiss Academy of Medical Sciences (SAMW), Bern, Switzerland. Boehringer Ingelheim, Astra Zeneca and Mundipharma also contributed with a financial support in this study.

# **ACKNOWLEDGMENTS**

Special thanks to the following institution and Departments for their support in recruitment of the study patients: Marketing Department (Cantonal Hospital Baselland, Liestal, Switzerland), Dr. med. A. Breitenbücher (pulmonologist, Cantonal Hospital Baselland, Bruderholz, Switzerland), Dr. med. L. Joos (pulmonologist, Claraspital, Basel, Switzerland), Dr. med. S. Vogt (pulmonologist, Hospital Rheinfelden, Rheinfelden, Switzerland), Dr. med. M. Frey (pulmonologist, Clinic Barmelweid, Barmelweid, Switzerland) and Dr. med. D. Simonett, privat practice pulmonologist, Liestal, Switzerland). The authors also acknowledge the efforts of Anna-Lisa Flamm, Research Nurse, who contributes with a lot of patience at the data collection.

# **COMPETING INTERESTS**

None declared.

# ETHICS APPROVAL

Ethics Committee of Nordwest- and Zentralschweiz (EK- 269/13).

# REFERENCES

- 1. Global suveillance, prevention and control of chronic respiratory diseases: a comprehensive approach. World Health Organization 2007. http://www.who.int/gard/publications/GARD%20Book%202007.pdf?ua=1 (accessed January 2017).
- 2. World Health Statistics. World Health Organization 2008. http://www.who.int/gho/publications/world\_health\_statistics/EN\_WHS08\_Full.pdf (accessed January 2017).
- 3. Lopez-Campos, JL, Tan W, Soriano JB. *Global burden of COPD.* Respirology, 2016;21(1):14-23.
- 4. Braman SS. *The global burden of asthma*. Chest, 2006;130(1 Suppl):4S-12S.
- 5. Wuthrich, B, Schmid-Grendelmeier P, Schindler C, et al. *Prevalence of atopy and respiratory allergic diseases in the elderly SAPALDIA population*. Int Arch Allergy Immunol, 2013;162(2):143-8.
- 6. Bridevaux PO, Probst-Hensch NM, Schindler C, et al. *Prevalence of airflow obstruction in smokers and never-smokers in Switzerland.* Eur Respir J, 2010;36(6):1259-69.
- 7. Jochmann A, Scherr A, Jochmann DC, et al. *Impact of adherence to the GOLD guidelines on symptom prevalence, lung function decline and exacerbation rate in the Swiss COPD cohort.* Swiss Med Wkly, 2012;142:w13567.
- 8. Soler-Cataluna JJ, Martinez-Garcia MA, Roman Sanchez P, et al. Severe acute exacerbations and mortality in patients with chronic obstructive pulmonary disease. Thorax, 2005;60(11):925-31.
- 9. Leuppi JD, Steurer-Stey C, Peter M, et al. *Asthma control in Switzerland: a general practitioner based survey.* Curr Med Res Opin, 2006;22(11):2159-66.
- 10. Miedinger D, Neukomm E, Chhajed PN, et al. *The use of the Asthma Control Test in general practice and its correlation with asthma control according to the GINA guidelines*. Curr Med Res Opin, 2011;27(12):2301-8.
- 11. Taegtmeyer AB, Steurer-Stey C, Price DB, et al. *Predictors of asthma control in everyday clinical practice in Switzerland*. Curr Med Res Opin, 2009;25(10):2549-55.
- 12. Leuppi JD. [Adherence to asthma therapy]. Ther Umsch, 2010;67(6): 323-7.
- 13. Adherence to long-term therapies: evidence for action. World Health Organization 2003. http://www.who.int/chp/knowledge/publications/adherence\_full\_report.pdf?ua=1 (accessed January 2017).
- 14. Heuer H, Heuer S, Lenneck K. *Compliance in der Arzneitherapie: Von der Non-Compliance zu pharmazeutischer und medizinischer Kooperation.* Wissenschaftliche Verlagsgesellschaft mbH Stuttgart, 1999.
- 15. Vrijens B, De Geest S, Hughes DA, et al. *A new taxonomy for describing and defining adherence to medications*. Br J Clin Pharmacol, 2012;73(5):691-705.
- 16. Haynes RB, Montague P, Oliver T, et al. *Interventions for helping patients to follow prescriptions for medications*. Cochrane Database Syst Rev, 2002(2);CD000011.
- 17. Osterberg L, Blaschke T. *Adherence to medication.* N Engl J Med, 2005;353(5):487-97.
- 18. Vrijens B, Dima AL, Van Ganse E, et al. What We Mean When We Talk About Adherence in Respiratory Medicine. J Allergy Clin Immunol Pract, 2016;4(5):802-12.
- 19. Lehmann A, Aslani P, Ahmed R, et al. *Assessing medication adherence: options to consider.* Int J Clin Pharm, 2014;36(1):55-69.
- 20. Sumino K, Cabana MD. *Medication adherence in asthma patients*. Curr Opin Pulm Med, 2013;19(1):49-53.
- 21. Sutton S, Kinmonth AL, Hardeman W et al, *Does electronic monitoring influence adherence to medication? Randomized controlled trial of measurement reactivity.* Ann Behav Med, 2014;48(3):293-9.

- 22. Makela MJ, Backer V, Hedegaard M, et al. *Adherence to inhaled therapies, health outcomes and costs in patients with asthma and COPD.* Respir Med, 2013;107(10):1481-90.
- 23. Krishnan JA, Bender BG, Wamboldt FS, et al. *Adherence to inhaled corticosteroids:* an ancillary study of the Childhood Asthma Management Program clinical trial. J Allergy Clin Immunol, 2012;129(1):112-8.
- 24. Feehan M, Ranker L, Durante R, et al. *Adherence to controller asthma medications:* 6-month prevalence across a US community pharmacy chain. J Clin Pharm Ther Published Online First: 20 August 2015. doi:10.1111/jcpt.12316.
- 25. Gamble J, Stevenson M, McClean E, et al. *The prevalence of nonadherence in difficult asthma*. Am J Respir Crit Care Med, 2009;180(9):817-22.
- 26. Jung E, Pickard AS, Salmon JW, et al. *Medication adherence and persistence in the last year of life in COPD patients*. Respir Med, 2009;103(4):525-34.
- 27. Steiner JF, Prochazka AV. *The assessment of refill compliance using pharmacy records: methods, validity, and applications.* J Clin Epidemiol, 1997;50(1):105-16.
- 28. Simmon MS, Nides MA, Kleerup EC, et al. *Validation of the Doser, a new device for monitoring metered-dose inhaler use.* J Allergy Clin Immunol, 1998;102(3):409-13.
- 29. Coutts JA, Gibson NA, Paton JY. *Measuring compliance with inhaled medication in asthma*. Arch Dis Child, 1992;67(3):332-3.
- 30. Burgess SW, Wilson SS, Cooper DM et al. *In vitro evaluation of an asthma dosing device: the smart-inhaler.* Respir Med, 2006;100(5):841-5.
- 31. Keemink YS, Klok T, Brand PL. Long-term adherence to daily controller medication in children with asthma: The role of outpatient clinic visits. Pediatr Pulmonol, 2015;50(11):1060-4.
- 32. Patel M, Pilcher J, Travers J, et al. *Use of metered-dose inhaler electronic monitoring in a real-world asthma randomized controlled trial.* J Allergy Clin Immunol Pract, 2013;1(1):83-91.
- 33. Charles T, Quinn D, Weatherall M, et al. *An audiovisual reminder function improves adherence with inhaled corticosteroid therapy in asthma*. J Allergy Clin Immunol, 2007;119(4):811-6.
- 34. Arnet I, Walter PN, Hersberger KE. *Polymedication Electronic Monitoring System (POEMS) a new technology for measuring adherence.* Front Pharmacol, 2013;4:26.
- 35. Haynes RB, Ackloo E, Sahota N, et al. *Interventions for enhancing medication adherence*. Cochrane Database Syst Rev, 2008(2):CD000011.
- 36. Richtig inhalieren. Deutsche Atemwegsliga e.V. In der Deutschen Gesellschaft für Pneumologie. http://www.atemwegsliga.de/richtig-inhalieren.html (accessed January 2017)
- 37. Melani AS, Zanchetta D, Barbato N, et al. *Inhalation technique and variables associated with misuse of conventional metered-dose inhalers and newer dry powder inhalers in experienced adults*. Ann Allergy Asthma Immunol, 2004;93(5):439-46.
- 38. Ronmark E, Jogi R, Lindqvist A, et al. *Correct use of three powder inhalers: comparison between Diskus, Turbuhaler, and Easyhaler.* J Asthma, 2005;42(3):173-8.
- 39. Nimmo CJ, Chen DN, Martinusen SM, et al. Assessment of patient acceptance and inhalation technique of a pressurized aerosol inhaler and two breath-actuated devices. Ann Pharmacother, 1993;27(7-8):922-7.
- 40. van der Palen J, Klein JJ, Kerkhoff AH et al. *Evaluation of the long-term effectiveness of three instruction modes for inhaling medicines*. Patient Educ Couns, 1997;32(1 Suppl):S87-95.
- 41. Jones PW, Harding G, Berry P, et al. *Development and first validation of the COPD Assessment Test.* Eur Respir J, 2009;34(3):648-54.
- 42. Nathan RA, Sorkness CA, Kosinski M, et al. *Development of the asthma control test: a survey for assessing asthma control.* J Allergy Clin Immunol, 2004;113(1):59-65.
- 43. Jones PW, Quirk FH, Baveystock CM. *The St George's Respiratory Questionnaire*. Respir Med, 1991;85 Suppl B:25-31; discussion 33-7.

- 44. Ware JE Jr, Sherbourne CD. *The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection.* Med Care, 1992;30(6):473-83.
- 45. Horne R, Weinman J. *Patients' beliefs about prescribed medicines and their role in adherence to treatment in chronic physical illness*. J Psychosom Res, 1999;47(6): 555-67.
- 46. Mahler C, Hermann K, Horne R, et al. *Patients' beliefs about medicines in a primary care setting in Germany.* J Eval Clin Pract, 2012;18(2):409-13.
- 47. Leuppi JD, Schuetz P, Bingisser R, et al. *Short-term vs conventional glucocorticoid therapy in acute exacerbations of chronic obstructive pulmonary disease: the REDUCE randomized clinical trial.* JAMA, 2013;309(21):2223-31.
- 48. Rodriguez-Roisin R. *Toward a consensus definition for COPD exacerbations.* Chest, 2000;117(5 Suppl 2): 398S-401S.
- 49. Eisen SA, Hanpeter JA, Kreuger LW, et al. *Monitoring medication compliance:* description of a new device. J Compliance Health Care, 1987;2(2):131-42.
- 50. Product information Onbrez, Novartis Pharma Schweiz AG, Rischi; Domizil 6343 Rotkreuz, Switzerland. Compendium (2014) http://compendium.ch/mpub/pnr/1154498/html/de#7900 (accessed January 2017).
- 51. Product information Seretide, GlaxoSmithkline AG Münchenbuchsee, Switzerland. Compendium (2014). http://compendium.ch/mpub/pnr/73528/html/de (accessed January 2017)
- 52. Product information Spiriva, Boehringer Ingelheim GmbH, 4002 Basel, Switzerland. Compendium (2012). http://compendium.ch/mpub/pnr/1009898/html/de (accessed January 2017).
- 53. Product information Symbicort, AstraZeneca Ag, Zug, Switzerland. Compendium (2016). http://compendium.ch/mpub/pnr/93069/html/de (accessed January 2017).
- 54. Product information Ventolin, GlaxoSmithkline AG Münchenbuchsee, Switzerland. Compendium (2007). http://compendium.ch/mpub/pnr/83981/html/de#7900 (accessed: January 2017).
- 55. Product information Relvar, GlaxoSmithKline AG Münchenbuchsee, Switzerland. Compendium (2016). http://compendium.ch/mpub/pnr/1258609/html/de#7900 (accessed January 2017).
- 56. White IR, Royston P. *Imputing missing covariate values for the Cox model.* Stat Med, 2009;28(15):1982-98.
- 57. Bourbeau J, Bartlett SJ, *Patient adherence in COPD.* Thorax, 2008;63(9): 831-8.
- 58. Lam WY, Fresco P. *Medication Adherence Measures: An Overview.* Biomed Res Int, 2015;2015:217047.

# LEGEND OF FIGURES

Figure 1: Study flow chart based on the CONSORT (Consolidated Standards of Reporting Trials) guidelines.